CLINICAL TRIAL: NCT04465825
Title: Developing Strategies to Optimize the Exercise Response in Persons Living With Tetraplegia.
Brief Title: Developing Strategies to Optimize the Exercise Response After Tetraplegia.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HS22987
Record Dates: First submitted 2020-07-07; First posted 2020-07-10 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2020-06

CONDITIONS: Spinal Cord Injuries; Spinal Cord Injury Cervical; Paraplegia, Spinal
Keywords: exercise
MeSH Terms: conditions — Spinal Cord Injuries; Paraplegia; Motor Activity

STUDY DESIGN:
Intervention Model Description: Part 2 is a randomized crossover design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interspersing HITT in exercise (Active Comparator): We will test whether introducing HITT into an acute exercise bout will increase overall energy expenditure or time to fatigue.
  Interventions: Behavioral: HITT: intermittent high intensity exercise
- Acute exercise bout with no HITT (No Intervention): Exercise will occur at 50% peak without introducing HITT.

INTERVENTIONS:
Behavioral: HITT: intermittent high intensity exercise — Intermittent bouts of 30-60 seconds of exercise at 90% of peak intensity (HITT).
  Arms: Interspersing HITT in exercise

SUMMARY:
To identify means to improve exercise performance in participants with tetraplegia.

DETAILED DESCRIPTION:
Part I. This study will examine the relationship between steady-state and peak exercise performance in participants with tetraplegia or paraplegia.

Participants will have their peak energy expenditure measured using a discontinuous step test. Participants will then perform three different trials of exercise at a steady state at a target intensity that corresponds with 90%, 70%, and 60% of their own measured peak energy expense. Participants will exercise at the prescribed power output until fatigue. Participants may choose which exercise mode they use (with all steady-state trials being in the same mode as the peak test), and may choose to perform the study twice in the different exercise modes. Exercise trials will be performed over a number of different sessions in a randomized order, allowing for adequate rest and recovery between trials, and depending on each participant's capabilities and preferences.

Part II. This study will determine if high intensity interval training (HIIT) results in greater energy expense than constant rate aerobic exercise, and will test if exercising with HITT effects time to fatigue.

Participants will exercise using a high intensity interval training (HIIT) protocol, which involves alternating high intensity bouts of short duration with low intensity bouts of longer duration. Participants will have their peak energy expenditure measured using a discontinuous step test. Participants will then perform one trial of steady-state exercise at a target intensity that corresponds with 50% of their peak energy expense, for a target of 20-45 minutes. Participants will perform a separate trial using a HIIT protocol of exercise at a target intensity that corresponds with 50% of their peak energy expense interspersed with bouts of high intensity (target intensity that corresponds with 90% of peak energy expense) for 30-60 seconds, for a total duration target of 20-45 minutes.

Participants may choose which exercise mode they use (with all trials being in the same mode as the peak test), and may choose to perform the study twice in the different exercise modes. Exercise trials will be performed over a number of different sessions in a randomized order, allowing for adequate rest and recovery between trials, and depending on each participant's capabilities and preferences.

ELIGIBILITY:
Inclusion Criteria:

* Spinal cord injury of at least one year duration, C5-T12, ASIA impairment scale (AIS) A-D
* Aged 18-75 years for the duration of the study participation
* Medically stable and healthy enough to engage in and complete exercise requirements
* Willing and able to complete the exercise protocols and testing requirements
* Able to understand and follow written and verbal instructions from study staff
* Able to communicate with study staff about their exercise capabilities and preferences

Exclusion Criteria:

* Current serious injury(ies) of the upper extremities
* Known cardiovascular disease
* Unsatisfactory results of EKG screening
* Implanted electronic cardiac device (e.g. pace maker, defibrillator, etc.)
* Current pressure ulcer(s)
* Morbid obesity
* Known thyroid dysfunction
* Current cancer
* Current uncontrolled high blood pressure ( > 140/90 mmHg)
* Uncontrolled epilepsy
* Current deep vein thrombosis
* Ventilator-dependent
* Cognitive impairment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2021-11 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Energy expenditure in ml of oxygen consumed per minute per kg of body weight | Measured during 20-40 minutes of exercise
  Estimation of energy expenditure for bout of exercise
Time to fatigue | Measured during 20-40 minutes of exercise
  Total duration of exercise

SECONDARY OUTCOMES:
Ratings of perceived exertion | Measured during 20-40 minutes of exercise
  Ratings of perceived exertion during exercise
Heart rate | Measured during 20-40 minutes of exercise
  We will examine differences in average, peak HR and HR variability

IPD SHARING:
Plan to Share IPD: Yes
Once published we will strive to make anonymized study data available.
Supporting Information: Study Protocol, ICF
Time Frame: The data will be available once published for one year.